CLINICAL TRIAL: NCT07285304
Title: A Phase 3 Long-term Study of TS-172 in Hyperphosphatemia Patients on Hemodialysis With Phosphate Binders
Brief Title: A Long-term Study of TS-172 in Hyperphosphatemia Patients on Hemodialysis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS172-03-03
Record Dates: First submitted 2025-11-24; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hyperphosphatemia Patients on Hemodialysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TS-172 (Experimental)
  Interventions: Drug: TS-172

INTERVENTIONS:
Drug: TS-172 — oral administration of TS-172 20~60 mg/day

SUMMARY:
A clinical study to evaluate the long-term safety and efficacy of TS-172 in hyperphosphatemia patients on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Hyperphosphatemia patients (outpatients) with chronic kidney disease receiving hemodialysis (HD or HDF) 3 times a week for at least 12 weeks prior to Visit 1 (Week -2)
2. Patients aged ≥18 years at the time of obtaining informed consent
3. Patients who have been prescribed at least one phosphate binder within the approved dosage, and the prescribed drug and dosage regimen should have been unchanged during the last 2 weeks prior to Visit 1 (Week -2)
4. Patients with a serum phosphorus concentration of ≥ 3.5 mg/dL and ≤ 7.0 mg/dL at Visit 1 (Week -2) or Visit 2 (Week -1)

Exclusion Criteria:

1. Patients with confirmed serum intact PTH concentration >500 pg/mL at Visit 1 (Week -2)
2. Patients who have undergone previous parathyroid intervention (PTx, PEIT, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 26 weeks or up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No